CLINICAL TRIAL: NCT02867514
Title: Evaluation de l'Effet de la Stimulation Transcranienne en Courant Continu Chez Les Personnes Tabagiques dépendantes
Brief Title: Effect of the Transcranial Direct Current Stimulation (tDCS) on Dependent Smoking People
Acronym: TabaSCo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P/2012/133
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Tobacco Abuse Smoke
Keywords: tobacco; craving; tDCS; attentional tasks
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- anodal tDCS on left DLPFC (F3) (Active Comparator): tDCS is a non-invasive neuromodulation method, which delivers a constant current of low intensity (1 mA) during 30 min for 10 sessions. Anode is placed on the scalp facing on left DLPFC and cathode on right DLPFC.
  Interventions: Device: transcranial Direct Current Stimulation (tDCS)
- sham tDCS on left DLPFC (F3) (Sham Comparator): tDCS differs from active tDCS by the interruption of stimulation after 15 sec and reactivation of the stimulation 15 sec before the end of the session (30 min - 10 sessions). Anode is placed on the scalp facing on left DLPFC and cathode on right DLPFC.
  Interventions: Device: transcranial Direct Current Stimulation (tDCS)
- anodal tDCS on right DLPFC (F4) (Active Comparator): tDCS is a non-invasive neuromodulation method, which delivers a constant current of low intensity (1 mA) during 30 min for 10 sessions. Anode is placed on the scalp facing on right DLPFC and cathode on left DLPFC.
  Interventions: Device: transcranial Direct Current Stimulation (tDCS)
- sham tDCS on right DLPFC (F4) (Sham Comparator): tDCS differs from active tDCS by the interruption of stimulation after 15 sec and reactivation of the stimulation 15 sec before the end of the session (30 min - 10 sessions). Anode is placed on the scalp facing on right DLPFC and cathode on left DLPFC.
  Interventions: Device: transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: transcranial Direct Current Stimulation (tDCS) — After locating the stimulation areas, treatment will be delivered during 30-minute session. Treatment will be occur 1 session per day during 10 days (5 days per week during 2 successive weeks). Subjects will be monitored during tDCS for any side effects or adverse events.
  Other Names: EldithDC-NeuroConn Stimulator (NeuroConn Gmbh, Germany)

SUMMARY:
The purpose of this study is to evaluate the effect of 10 sessions of anodal transcranial Direct Current Stimulation (tDCS - 1 mA) applied to left vs right CDLPF of tobacco-dependent subjects compared to the application of a placebo tDCS (sham procedure) on the craving, which is evaluated by the item 1 of Fagerström test between day 1 and day 10. Craving is also evaluated 1 month post-treatment.

DETAILED DESCRIPTION:
Tobacco is the second leading cause of death worldwide. It is currently responsible for the death of one in 10 adults (about 5 million deaths per year) and it is the fourth disease risk factor in the world. Many methods to quit smoking are available but in all cases, relapse is a common phenomena. The main risk factor for relapse is craving. So, acting on the craving seems essential to modulate tobacco consumption. Many functional neuroimaging studies have established a neuroanatomical substrate for craving process, in particularly dorsolateral prefrontal cortex (DLPFC), accessible par neuromodulation.

ELIGIBILITY:
Inclusion Criteria:

* Fagerström score ≥ 5
* Q-MAT score ≥ 6
* smoking subjects from 10 to 30 cigarettes a day
* right-handed subjects
* w/o severe progressive somatic pathology (especially tumor diseases, degenerative diseases)
* Hamilton Depression Rating Scale-17 score <18

Exclusion Criteria:

* pregnancy and/or lactation
* presence of a specific contraindication for tDCS (e.g. personal history of epilepsy, metallic head implant, cardiac pacemaker...)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-03; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
change from baseline in craving evaluated by item 1 of Fagerström test | baseline, day 10 and 1 month post-ttt
  before and after the 10 sessions

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Haffen, Prof, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (2):
- France (2):
  - CHRU Besancon - Service de Psychiatrie - Centre Investigation Clinique Innovation Technologique (CIC-IT808), Besançon
  - Assistance Publique - Hôpitaux de Paris, Paris

IPD SHARING:
Plan to Share IPD: No